CLINICAL TRIAL: NCT03519607
Title: The Impact of a Self-help Coping App on Distress Levels in Men Experiencing Infertility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fertility Centers of Illinois (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20180901
Record Dates: First submitted 2018-04-06; First posted 2018-05-09 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Stress Reduction
Keywords: Infertility; Distress; Coping; Men
MeSH Terms: conditions — Infertility; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Intervention Model Description: Comparison of distress scores between the intervention group and the control group
Who Masked: Outcomes Assessor
Masking Description: Participant assignment will be masked for data analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Active Comparator): Participants who are in the intervention group will receive the FertiStrong app downloading instructions as soon as they have been randomized. They will have access to this app for a period of 30 days during the intervention phase of the study.
  Interventions: Behavioral: FertiStrong App
- Control Group (No Intervention): Participants in the control group will not have access to the FertiStrong app for the first 30 days. After a period of 30 days, participants will be provided downloading instructions to this app.

INTERVENTIONS:
Behavioral: FertiStrong App — The FertiStrong mobile app is similar to FertiCalm, which is designed for women with infertility. FertiCalm (www.FertiCalm.com) can be downloaded for free anywhere in the US, for both Apple and Android phones. Each app contains twelve main categories and each main category contains up to five tailored situations. For each situation, there are six options. Three of the options are the same for all situations (humor, self-nurture, relaxation) and three are unique (cognitive solutions, behavioral solutions, social solutions).
  Other Names: FertiStrong
  Arms: Treatment Group

SUMMARY:
The purpose of this study is to determine if the use of a new app, FertiStrong, is associated with decreased levels of anxiety and depression in men who have infertility or whose partner has infertility.

DETAILED DESCRIPTION:
Individuals who are experiencing infertility report high levels of anxiety and depression. A recent study (1) documented that both men and women involved in the treatment of infertility expressed emotional distress. Research on the female partner of an infertile couple documents that psychological interventions, especially those with a cognitive-behavior therapy (CBT) focus, are associated with significant decreases in levels of anxiety and depression (2). Subsequent research has also shown that both members of the infertile couple definitively underutilize the psychological services offered to them. Thus, new ways to provide psychological relief to these individuals is needed. This has lead to the development of a new app, FertiStrong. This app is targeted at men- either men with infertility or men whose partner has infertility.

Study Requirements:

1. Study participants will be asked to complete an on-line questionnaire.
2. Once completed, the study participant will be randomly assigned to one of two groups. One group will be provided the mobile app to use for 30 days. The second group will be provided the app after 30 days.
3. After the 30 day period, each group will be asked to complete a follow-up questionnaire. Each questionnaire will take approximately 15-20 minutes to compete.

Men who are directly seeking care or whose partners is seeking care at any Fertility Center of Illinois location are invited to participate.

ELIGIBILITY:
Inclusion Criteria:

* All men who are receiving care, or whose partner is receiving care, at Fertility Centers of Illinois during the study period.

Exclusion Criteria:

1. Does not have daily access to a smart phone
2. Does not read or understand English

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Males experiencing infertility, or men whose partner is experiencing infertility
Enrollment: 100 (Estimated)
Dates: Start 2018-04-30 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety and Depression in Men Experiencing Infertility | 6 months post study completion
  Evaluation of pre and post Hospital Anxiety and Depression Scores

SECONDARY OUTCOMES:
Stress Levels in Men Experiencing Infertility | 6 months post study completion
  Fertility related distress will be measured using the Fertility Problem inventory (FPI)

CONTACTS AND LOCATIONS:
Overall Officials: Meike Uhler, MD, Principal Investigator — Fertility Centers of Illinois
Locations (1):
- Fertility Centers of Illinois, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No